CLINICAL TRIAL: NCT00031889
Title: A Randomized Phase II Trial of Exemestane With and Without Bicalutamide as Second Line Therapy After Failure of Androgen Suppression in Advanced Prostate Cancer
Brief Title: Exemestane With or Without Bicalutamide in Treating Patients With Stage IV Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 09/01; EU-20139
Record Dates: First submitted 2002-03-08; First posted 2003-07-01 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oral exemestane once daily
  Interventions: Drug: Exemestane
- Arm II (Active Comparator): Patients receive exemestane as in arm I and oral bicalutamide once daily
  Interventions: Drug: Exemestane+bicalutamide

INTERVENTIONS:
Drug: Exemestane — Exemestane
  Arms: Arm I
Drug: Exemestane+bicalutamide — Exemestane as in arm I and oral bicalutamide once daily
  Arms: Arm II

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using exemestane plus bicalutamide may fight prostate cancer by reducing the production of androgens. It is not yet known if exemestane is more effective with or without bicalutamide in treating prostate cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of exemestane with or without bicalutamide in treating patients who have stage IV prostate cancer that has been previously treated with hormone therapy or surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy and tolerability of exemestane with or without bicalutamide as second-line therapy after failure of androgen suppression (luteinizing hormone-releasing hormone agonist or orchiectomy) in patients with stage IV prostate cancer.
* Determine the potential antagonistic effect of the weak androgen action of exemestane when combined with bicalutamide in these patients.
* Compare the quality of life (QOL) in patients treated with these regimens.
* Correlate prostate-specific antigen response and data of QOL, including scores for pain intensity and analgesic consumption, in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (0 vs 1-2), pain (none or mild vs moderate or severe), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral exemestane once daily.
* Arm II: Patients receive exemestane as in arm I and oral bicalutamide once daily.

Treatment in both arms continues every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

Quality of life and pain are assessed at baseline, on day 1 of course 2 and any subsequent courses, and at disease progression or treatment failure (if applicable).

Patients are followed monthly until disease progression.

PROJECTED ACCRUAL: A total of 20-62 patients (10-31 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV adenocarcinoma of the prostate
* Documented disease progression based on prostate-specific antigen (PSA) progression during first-line androgen suppression (luteinizing hormone-releasing hormone agonist or orchiectomy)

  * PSA progression is defined by the following:

    * Interval of at least 1 week between reference value (time point value 1) and the next PSA level (time point value 2)
    * PSA at time point value 3 is greater than PSA at time point value 2 OR
    * PSA at time point value 3 is not greater than PSA at time point value 2, but PSA at time point value 4 is greater than PSA at time point value 2
* PSA at least 5 ng/mL
* Must continue primary androgen suppression if no prior surgical castration
* No known leptomeningeal or brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No acute concurrent severe infection
* No other concurrent significant disease that would preclude study therapy
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior antibody or gene therapy

Chemotherapy:

* No prior cytostatic agents

Endocrine therapy:

* See Disease Characteristics
* No prior estramustine
* No prior antiandrogens (e.g., bicalutamide)
* No concurrent estrogen-containing medicine

Radiotherapy:

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy to more than 1 field

Surgery:

* See Disease Characteristics

Other:

* At least 4 weeks since prior investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2001-08; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bonomo, MD, Study Chair — Ospedale Beata Vergine
Locations (12):
- Switzerland (12):
  - Kantonspital Aarau, Aarau
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Ratisches Kantons und Regionalspital, Chur
  - Clinique De Genolier, Genolier
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Ospedale Beata Vergine, Mendrisio
  - Institut Central des Hopitaux Valaisans, Sion
  - Universitaetsspital, Zurich